CLINICAL TRIAL: NCT02685709
Title: A Phase 3, Randomized, Active Controlled Study to Evaluate Maintenance of Response, Safety and Patient Reported Outcomes in Acromegaly Patients Treated With Octreotide Capsules vs. Parenteral Somatostatin Receptor Ligands
Brief Title: Comparison of Oral Octreotide Capsules to Injectable Somatostatin Analogs in Acromegaly
Acronym: MPOWERED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiasma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OOC-ACM-302; 2015-002854-11 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-19 (Estimated); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Acromegaly
Keywords: Octreotide Capsules; Acromegaly; somatostatin receptor ligands (SRLs); Mpowered; OOC-ACM-302
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Run-in phase (Experimental): Oral octreotide capsules
  Interventions: Drug: Octreotide capsules
- RCT phase - Oral (Experimental): Oral octreotide capsules
  Interventions: Drug: Octreotide capsules
- RCT phase - Injectables (Active Comparator): Injectable somatostatin analogs (octreotide or lanreotide)
  Interventions: Drug: Octreotide capsules
- Combination phase (sub-study) (Experimental): Octreotide capsules plus cabergoline
  Interventions: Drug: Octreotide capsules

INTERVENTIONS:
Drug: Octreotide capsules
  Other Names: Injection SRLs

SUMMARY:
Octreotide capsule is a novel, orally-administered formulation of the commercially-available injectable drug octreotide. In a recent phase 3 trial (OPTMAL; NCT03252353), oral octreotide capsules demonstrated sustained biochemical response up to 13 months in patients with acromegaly previously managed with somatostatin analog injections (ref).

The objective of this study was to compare the efficacy, safety, and patient reported outcomes (PROs) between oral octreotide capsules and injectable somatostatin receptor ligands (SRLs).

DETAILED DESCRIPTION:
This was phase 3, randomized, open-label, active controlled, multicenter study to evaluate the maintenance of response, safety and patient reported outcomes (PROs) in acromegaly patients treated with octreotide capsules and in patients treated with standard of care parenteral somatostatin receptor ligands (SRLs), who previously tolerated and demonstrated biochemical control on both treatments.

The core study consisted of three phases: a Screening phase, Run-in phase and a Randomized Controlled Treatment (RCT) phase.

Eligible patients who were biochemically controlled on parenteral SRLs were switched to octreotide capsules for a 26-week period Run-in phase. During this phase the effective dose for each patient was determined through dose titration.

Patients whose acromegaly has been controlled biochemically on octreotide capsules at the end of the Run-in phase entered a 36-week open-label RCT phase, where they randomized to continue on octreotide capsules or switch back to their injectable SRL treatment (as received prior to Screening).

Following the completion of the core study (Screening, Run-in and RCT phases), eligible patients were offered to enter the Study Extension phase and receive octreotide capsules until product marketing or study termination.

A Sub-study, performed in selected non-European sites, allowed patients with inadequate biochemical control on octreotide capsules during the Run-in phase to enter a Combination phase and receive co-administration of octreotide capsules with cabergoline tablets for a total of 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acromegaly
* Treatment with Somatostatin analogs injections (octreotide or lanreotide) for at least 6 months
* Biochemical control (IGF -1 < 1.3 x ULN and GH < 2.5ng/mL)

Exclusion Criteria:

* Injections of long-acting somatostatin analogs, at a dosing interval > 8 weeks.
* Pituitary radiotherapy within 5 years
* Pituitary surgery within six months
* Patients who previously participated in CH-ACM-01 study
* Any clinically significant uncontrolled concomitant disease
* Symptomatic cholelithiasis
* Previous treatment with:
* Pegvisomant, within 12 weeks
* Dopamine agonists, within 6 weeks
* Pasireotide, within 12 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fleseriu, M.D., FACE, Study Chair — Northwest Pituitary Center, Oregon Health & Science University , Portland, OR, USA
Locations (53):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Keck Medical Center of University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas
- Austria (2):
  - Universitätsklinik für Innere Medizin Klinische Abteilung für Endokrinologie und Diabetologie, Graz
  - Medizinische Universität Wien, Vienna
- France (2):
  - Hospices Civils de Lyon, Bron
  - Hôpital Bicêtre APHP, Le Kremlin-Bicêtre
- Praxis für Endokrinologie und Diabetologie Dr M Droste, Oldenburg, Germany
- Hungary (3):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - University of Pecs, Pécs
  - Szegedi Tudományegyetem, I. Belgyógyászati Klinika, Szeged
- Italy (3):
  - Policlinico di Monserrato U.O.C. Endocrinologia e Diabetologia, Monserrato
  - Università di Pisa Dipartimento di Medicina Clinica e Sperimentale, Pisa
  - Fondazione Policlinico Universitario A. Gemelli Università Cattolica del S.Cuore S.C. Endocrinologia e Malattie del Metabolismo, Rome
- Lithuania (2):
  - Hospital of LUHS Kauno Klinikos, Kaunas
  - Vaidotas Urbanavicius Individuali Imonė, Vilnius
- Poland (2):
  - Katedra i Klinika Endokrynologii i Chorob Wewnetrznych Gdanski Uniwersytet Medyczny, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Klinika Endokrynologii, Diabetologii i Leczenia Izotopami, Wroclaw
- "C.I. Parhon" National Institute of Endocrinology I Clinical Endocrinology Department - Endemic goitier and its complications, Bucharest, Romania
- Russia (9):
  - Antrium Multidisciplinary Medical Clinic, Barnaul
  - Interregional Clinical Diagnostic Center, Kazan'
  - Regional State Budgetary Healthcare Institution Regional State Hospital, Krasnoyarsk
  - Sechenov Moscow First State Medical University, Moscow
  - "Atlas" Medical Center, Moscow
  - Vladimirsky Moscow Regional Research Clinical Institute, Moscow
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Federal State Budgetary Institution "V. A. Almazov Federal North-West Medical Research Centre" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - "Centre Diabetes" LLC, Samara
- Clinical Centre of Serbia, Clinic for Endocrinology Diabetes and Metabolic Diseases, Belgrade, Serbia
- Spain (5):
  - Hospital Universitario de la Ribera, Alzira
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
  - Campus Del Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester Royal Infirmary, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melmed S, Popovic V, Bidlingmaier M, Mercado M, van der Lely AJ, Biermasz N, Bolanowski M, Coculescu M, Schopohl J, Racz K, Glaser B, Goth M, Greenman Y, Trainer P, Mezosi E, Shimon I, Giustina A, Korbonits M, Bronstein MD, Kleinberg D, Teichman S, Gliko-Kabir I, Mamluk R, Haviv A, Strasburger C. Safety and efficacy of oral octreotide in acromegaly: results of a multicenter phase III trial. J Clin Endocrinol Metab. 2015 Apr;100(4):1699-708. doi: 10.1210/jc.2014-4113. Epub 2015 Feb 9. PMID 25664604
- [Background] Melmed S. New therapeutic agents for acromegaly. Nat Rev Endocrinol. 2016 Feb;12(2):90-8. doi: 10.1038/nrendo.2015.196. Epub 2015 Nov 27. PMID 26610414
- [Derived] Fleseriu M, Dreval A, Bondar I, Vagapova G, Macut D, Pokramovich YG, Molitch ME, Leonova N, Raverot G, Grineva E, Poteshkin YE, Gilgun-Sherki Y, Ludlam WH, Patou G, Haviv A, Gordon MB, Biermasz NR, Melmed S, Strasburger CJ. Maintenance of response to oral octreotide compared with injectable somatostatin receptor ligands in patients with acromegaly: a phase 3, multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2022 Feb;10(2):102-111. doi: 10.1016/S2213-8587(21)00296-5. Epub 2021 Dec 22. PMID 34953531
- See also: Click here for more information about Chiasma — http://www.chiasmapharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 146 patients were enrolled into the Run-in phase. A total of 116 patients completed the Run-in phase and 30 patients discontinued the Run in phase.
  Of the 116 patients who completed the Run-in phase, 92 patients with IGF-1<1.3 ULN entered the RCT phase, 11 patients with IGF-1≥1.3 and <2 ULN on the highest octreotide dose entered the Combination phase, and 13 patients did not continue treatment.
Pre-assignment Details: Prior to Run-in - all patients treated with SRLs (59.6% octreotide and 39.4% on lanreotide). 78.8% of patients were treated with medium to high doses of SRLs.
  Prior to RCT - all patients were on oral octreotide capsules.
Groups:
- Run-in Phase: Oral octreotide capsules
  Octreotide capsules: Octreotide capsules 40mg/day, 60mg/day, 80mg/day determined by individual dose titration
- RCT Phase - Oral: Oral octreotide capsules
  Octreotide capsules: Octreotide capsules 40mg/day, 60mg/day, 80mg/day
- RCT Phase - Injectables: Injectable somatostatin analogs (octreotide or lanreotide)
  Injectable Somatostatin Analogs (octreotide or lanreotide):
  Octreotide- 10, 20, 30, 40 mg. Lanreotide- 60, 90, 120mg.
- Combination Phase (Sub-study): Octreotide capsules plus cabergoline
  Octreotide capsules: Octreotide capsules 40mg/day, 60mg/day, 80mg/day
  Cabergoline: Cabergoline - Up to 3.5mg/week
Period: Run-in Phase
Arm/Group | Run-in Phase | RCT Phase - Oral | RCT Phase - Injectables | Combination Phase (Sub-study)
Started | 146 | 0 | 0 | 0
Completed | 116 (30 patients early terminated the Run-in phase and 24 patient were not randomized to RCT) | 0 | 0 | 0
Not Completed | 30 | 0 | 0 | 0
Period: RCT Phase
Arm/Group | Run-in Phase | RCT Phase - Oral | RCT Phase - Injectables | Combination Phase (Sub-study)
Started | 0 (116 patients completed the Run-in phase, out of which 92 were randomized to the RCT phase, and 24 were not randomized to the RCT phase. Out of these 24, 11 patients eneterd the combination phase.) | 55 | 37 | 0
Completed | 0 | 54 | 35 | 0
Not Completed | 0 | 1 | 2 | 0
Period: Combination Phase
Arm/Group | Run-in Phase | RCT Phase - Oral | RCT Phase - Injectables | Combination Phase (Sub-study)
Started | 0 | 0 | 0 | 14 (14 patients entered the combination phase (3 patients early discontinued the Run-in phase, and 11 patients completed Run-in and were not eligible to RCT phase).)
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Acromegaly patients who previously tolerated and demonstrated a biochemical control on SRLs
Groups:
- Run-in Phase; RCT Phase - Oral: Oral octreotide capsules
  Octreotide capsules: Octreotide capsules 40mg/day, 60mg/day, 80mg/day
- RCT Phase - Injectables: Injectable somatostatin analogs (octreotide or lanreotide)
  Injectable Somatostatin Analogs (octreotide or lanreotide): Octreotide - 10, 20, 30mg. Lanreotide 60,90, 120mg.
- Combination Phase (Sub-study): Octreotide capsules plus cabergoline
  Octreotide capsules: Octreotide capsules 40mg/day, 60mg/day, 80mg/day
  Cabergoline: Cabergoline - 3.5mg/week
- Total: Total of all reporting groups
Arm/Group | Run-in Phase | RCT Phase - Oral | RCT Phase - Injectables | Combination Phase (Sub-study) | Total
Number analyzed (Participants) | 146 | 55 | 37 | 14 | 252
Age, Categorical [Count of Participants; unit: Participants] — Population: Number of participants was breakdown per study phase.
  Participants
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase: <=18 years | 0 | 0 | 0 | 0 | 0
    Run-in phase: Between 18 and 65 years | 124 | 0 | 0 | 0 | 124
    Run-in phase: >=65 years | 22 | 0 | 0 | 0 | 22
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase: <=18 years | 0 | 0 | 0 | 0 | 0
    RCT phase: Between 18 and 65 years | 0 | 46 | 32 | 0 | 78
    RCT phase: >=65 years | 0 | 9 | 5 | 0 | 14
    Combination Phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination Phase: <=18 years | 0 | 0 | 0 | 0 | 0
    Combination Phase: Between 18 and 65 years | 0 | 0 | 0 | 11 | 11
    Combination Phase: >=65 years | 0 | 0 | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number of participants was breakdown per study phase.
  years
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase | 54.1 (10.5) |  |  |  | 54.1 (10.5)
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase |  | 54.1 (10.88) | 55.2 (8.78) |  | 54.5 (10.05)
    Combination phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase |  |  |  | 59.8 (5.82) | 59.8 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number of participants was breakdown per study phase.
  Participants
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase: Female | 94 | 0 | 0 | 0 | 94
    Run-in phase: Male | 52 | 0 | 0 | 0 | 52
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase: Female | 0 | 35 | 26 | 0 | 61
    RCT phase: Male | 0 | 20 | 11 | 0 | 31
    Combination phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase: Female | 0 | 0 | 0 | 10 | 10
    Combination phase: Male | 0 | 0 | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number of participants was breakdown per study phase.
  Participants
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase: Hispanic or Latino | 5 | 0 | 0 | 0 | 5
    Run-in phase: Not Hispanic or Latino | 130 | 0 | 0 | 0 | 130
    Run-in phase: Unknown or Not Reported | 11 | 0 | 0 | 0 | 11
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase: Hispanic or Latino | 0 | 1 | 2 | 0 | 3
    RCT phase: Not Hispanic or Latino | 0 | 50 | 33 | 0 | 83
    RCT phase: Unknown or Not Reported | 0 | 4 | 2 | 0 | 6
    Combination phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase: Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Combination phase: Not Hispanic or Latino | 0 | 0 | 0 | 14 | 14
    Combination phase: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number of participants was breakdown per study phase.
  Participants
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Run-in phase: Asian | 1 | 0 | 0 | 0 | 1
    Run-in phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Run-in phase: Black or African American | 3 | 0 | 0 | 0 | 3
    Run-in phase: White | 133 | 0 | 0 | 0 | 133
    Run-in phase: More than one race | 9 | 0 | 0 | 0 | 9
    Run-in phase: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    RCT phase: Asian | 0 | 0 | 0 | 0 | 0
    RCT phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    RCT phase: Black or African American | 0 | 2 | 0 | 0 | 2
    RCT phase: White | 0 | 49 | 35 | 0 | 84
    RCT phase: More than one race | 0 | 4 | 2 | 0 | 6
    RCT phase: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    Combination phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Combination phase: Asian | 0 | 0 | 0 | 0 | 0
    Combination phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Combination phase: Black or African American | 0 | 0 | 0 | 0 | 0
    Combination phase: White | 0 | 0 | 0 | 14 | 14
    Combination phase: More than one race | 0 | 0 | 0 | 0 | 0
    Combination phase: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Region of enrollment in the Run-in phase. Population: Region of enrollment was summarized in the Run-in phase only, where 146 were randomized.
  Participants
    Hungary: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Hungary | 3 |  |  |  | 3
    United States: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    United States | 37 |  |  |  | 37
    Spain: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Spain | 6 |  |  |  | 6
    Russia: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Russia | 65 |  |  |  | 65
    Austria: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Austria | 6 |  |  |  | 6
    Italy: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Italy | 2 |  |  |  | 2
    France: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    France | 10 |  |  |  | 10
    Lithuania: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Lithuania | 8 |  |  |  | 8
    Serbia: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Serbia | 8 |  |  |  | 8
    Germany: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Germany | 1 |  |  |  | 1
Region of Enrollment [Count of Participants; unit: Participants] — Region of enrollment in the RCT phase. Population: Region of enrollment was captured for the RCT phase only, where patients were randomized to either oral octreotide (55) or injectable SRLs (37) .
  Participants
    Hungary: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    Hungary |  | 1 | 1 |  | 2
    United States: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    United States |  | 14 | 10 |  | 24
    Spain: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    Spain |  | 1 | 3 |  | 4
    Russia: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    Russia |  | 24 | 18 |  | 42
    Austria: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    Austria |  | 5 | 0 |  | 5
    Italy: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    Italy |  | 1 | 0 |  | 1
    France: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    France |  | 4 | 2 |  | 6
    Lithuania: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    Lithuania |  | 1 | 1 |  | 2
    Serbia: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    Serbia |  | 4 | 2 |  | 6
Region of Enrollment [Count of Participants; unit: Participants] — Region of enrollment- Combination phase Population: Region of enrollment was only captured for the Combination phase sub-study, in which 14 patients were included. .
  Participants
    United States: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    United States |  |  |  | 3 | 3
    Russia: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Russia |  |  |  | 10 | 10
    Serbia: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Serbia |  |  |  | 1 | 1
IGF-1 levels [Mean (Standard Deviation); unit: X Upper limit of normal (ULN)] — IGF-1 levels normalized for age and gender. The upper limit of normal is 1.0 x ULN Population: Mean calculated is phase-specific.
  X Upper limit of normal (ULN)
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase | 0.9 (0.27) |  |  |  | 0.9 (0.27)
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase |  | 0.9 (0.35) | 0.8 (0.21) |  | 0.9 (0.30)
    Combination phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase |  |  |  | 1.5 (0.35) | 1.5 (0.35)
IGF-I categorical [Count of Participants; unit: Participants] — Population: Number calculated is phase-specific.
  Participants
    Run-in phase- ≤ 1 ULN: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase- ≤ 1 ULN | 98 | 0 | 0 | 0 | 98
    Run-in phase- > 1 to < 1.3 ULN: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase- > 1 to < 1.3 ULN | 38 | 0 | 0 | 0 | 38
    Run-in phase- ≥ 1.3 ULN: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase- ≥ 1.3 ULN | 10 | 0 | 0 | 0 | 10
    RCT phase- ≤ 1 ULN: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase- ≤ 1 ULN | 0 | 37 | 29 | 0 | 66
    RCT phase- > 1 to < 1.3 ULN: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase- > 1 to < 1.3 ULN | 0 | 12 | 8 | 0 | 20
    RCT phase- ≥ 1.3 ULN: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase- ≥ 1.3 ULN | 0 | 6 | 0 | 0 | 6
    Combination phase- ≤ 1 ULN: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase- ≤ 1 ULN | 0 | 0 | 0 | 1 | 1
    Combination phase- > 1 to < 1.3 ULN: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase- > 1 to < 1.3 ULN | 0 | 0 | 0 | 4 | 4
    Combination phase- ≥ 1.3 ULN: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase- ≥ 1.3 ULN | 0 | 0 | 0 | 9 | 9
GH [Mean (Standard Deviation); unit: ng/ mL] — Population: Data analyzed in study-specific.
  ng/ mL
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase | 0.88 (0.818) |  |  |  | 0.88 (0.818)
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase |  | 0.55 (0.544) | 0.62 (0.634) |  | 0.58 (0.579)
    Combination phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase |  |  |  | 0.94 (0.544) | 0.94 (0.544)
Acromegaly Index of Severity (AIS) symptom score [Mean (Standard Deviation); unit: units on a scale] — The Acromegaly Index of Severity (AIS) symptom score is calculated based on the presence and severity of 5 acromegaly signs/symptoms: headache, swelling of extremities, joint pain, sweating, and fatigue. Each symptom was graded from no symptoms (score 0), to mild symptoms (1), moderate (2), or severe symptoms (3). The minimal total score is 0 and the maximal is 15. Population: Analysis performed is phase-specific.
  units on a scale
    Run-in phase: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
    Run-in phase | 4.8 (3.1) |  |  |  | 4.8 (3.1)
    RCT phase: number analyzed (Participants) | 0 | 55 | 37 | 0 | 92
    RCT phase |  | 4.2 (2.92) | 5 (2.98) |  | 4.5 (2.96)
    Combination phase: number analyzed (Participants) | 0 | 0 | 0 | 14 | 14
    Combination phase |  |  |  | 6.8 (3.95) | 6.8 (3.95)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Are Biochemically Controlled Throughout the RCT Phase
Description: Proportion of patients who are biochemically controlled throughout the RCT phase. A patient was considered biochemically controlled if IGF-1 Time Weighted Average (TWA) during the RCT phase is <1.3 ULN
Time Frame: 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
Participants | 50 | 37
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; Test type: Non-Inferiority — An assessment of NI was made by comparing the lower bound of the two-sided 95% confidence interval (CI) for the difference in biochemical control (octreotide capsules - SRLs) to a NI margin of -20%; Stratified Miettinen & Nurminen (M&N); 95% CI Stratified Miettinen & Nurminen = -19.9, 95% CI 2-sided [-19.9 to 0.5]

2. Secondary Outcome: Proportion of Patients With Clinical and Biochemical Control at the End of the RCT Phase
Description: Proportion of patients with clinical and biochemical control at the end of the RCT phase. Patients were considered biochemically and clinically controlled if they met both of the following criteria:
  * Their IGF-1 TWA during the RCT phase was <1.3 times ULN
  * Their AIS score at week 62/EOT was maintained or reduced compared to week 26 (start of RCT phase)
Time Frame: Week 62/ End of treatment; EOT
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
Participants | 36 | 27
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; Secondary endpoints were analyzed without adjustment for multiplicity or predefined noninferiority margins and therefore were interpreted as exploratory. This endpoint is descriptive with no formal statistical hypothesis testing; Test type: Other; The statistical analysis was based on the stratified Miettinen & Nurminen (M&N) method

3. Secondary Outcome: Proportion of Patients Who Maintain or Reduce the Overall Number of Active Acromegaly Symptoms at the End of the RCT Phase
Description: Proportion of patients who maintain or reduce the overall number of active acromegaly symptoms at the end of the RCT phase (week 62/ EOT) , compared to week 26 (start of the RCT phase
Time Frame: 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
Participants | 41 | 26
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; [analysis description as in outcome 2, analysis 1]; Test type: Other; Clopper-Pearson method; The statistical analysis was based on the stratified Miettinen & Nurminen (M&N) method

4. Secondary Outcome: Proportion of Patients Who Maintain or Improve Their Overall Acromegaly Index of Severity (AIS) Score at the End of the RCT Phase
Description: Proportion of patients who maintain or improve their overall Acromegaly index of severity (AIS) score at the end of the RCT phase (improvement defined as a reduction of at least one point in the AIS score), compared to week 26 (start of the RCT phase)
Time Frame: 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
Participants | 40 | 25
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; [analysis description as in outcome 2, analysis 1]; Test type: Other; Confidence interval was applied; The statistical analysis was based on the stratified Miettinen & Nurminen (M&N) method

5. Secondary Outcome: Proportion of Patients of Those Completing the RCT Phase Who Entered the Study Extension Phase
Description: Proportion of patients of those completing the RCT phase (at a time octreotide capsules were not commercially available at the specific country), who entered the Study Extension phase, overall and by treatment group
Time Frame: 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 54 | 35
Participants | 34 | 18
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; Secondary endpoints were analyzed without adjustment for multiplicity or predefined noninferiority margins and therefore were interpreted as exploratory; Test type: Other; Clopper-Pearson method; Based on this analysis 63.0% of patients in the octreotide capsule group and 51.4% of patients in the SRL injection group entered the Study Extension phase

6. Secondary Outcome: Change in IGF-1 Levels in the RCT Phase
Description: Change in IGF-1 levels from the start of the randomized phase to the end of RCT phase.
  Complete Responder (CR) is defined as IGF-1 ≤ 1 x ULN; Partial Responder (PR) is defined as 1 x ULN < IGF-1 < 1.3 x ULN, and Non-Responder (NR): IGF-1 ≥ 1.3 x ULN
Time Frame: Change from Week 26 to week 62
Measure: Mean (Standard Deviation); unit: x Upper limit of normal ("ULN")
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
x Upper limit of normal ("ULN") | -0.01 (0.199) | -0.04 (0.133)
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; [analysis description as in outcome 2, analysis 1]; Test type: Other; The mean change in IGF-1 from RCT Baseline to the end of the RCT phase was calculated using the Last Observation Carried Forward (LOCF) approach

7. Secondary Outcome: Change in GH Levels in the RCT Phase
Description: Change in GH levels from the start of the randomized phase through the end of RCT phase.
Time Frame: Change from Week 26 to week 62
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
ng/mL | -0.02 (0.506) | 0.27 (1.219)
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; [analysis description as in outcome 2, analysis 1]; Test type: Other; Estimates were obtained from an analysis of covariance (ANCOVA) for the mean integrated growth hormone (GH) change from baseline with explanatory factors of treatment group and baseline value

8. Other Pre Specified Outcome: Proportion of Patients Reporting Injection Site Reactions in the Acro-TSQ During the RCT Phase
Description: Proportion of patients reporting injection site reactions (ISRs). Acromegaly treatment satisfaction questionnaire (ACRO-TSQ) is a validated PRO tool assessing overall convenience and satisfaction with treatment and patient perception of symptomatic control and adverse drug. It includes 6 scales: Symptom Interference, (4 items); Treatment Convenience, (6 items); Injection Site Interference (2 items); GI Interference (3 items); Treatment Satisfaction, (3 items); and Emotional Reaction (3 items). Each scale score can range from 0 to 100, with 0 representing the lowest (highest burden/lower satisfaction) and 100 representing the best possible score (lowest burden/highest satisfaction) for each of the 6 scales. Positive ACRO-TSQ change scores indicate improvement while negative change scores indicate worsening.
Time Frame: 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 36
Participants | 0 | 17
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; This endpoint is descriptive with no formal statistical hypothesis testing; Test type: Other; The week 26 value was used as the baseline value for the RCT phase. The denominator for the percentage was the number of subjects at each visit

9. Other Pre Specified Outcome: Proportion of Patients Reporting Interference With Daily Activities in Acro-TSQ During the RCT Phase
Description: Proportion of patients reporting interference with daily activities in the Acromegaly Treatment Satisfaction Questionnaire (Acro-TSQ) during the RCT phase.
  Acro-TSQ is a validated PRO tool assessing overall convenience and satisfaction with treatment and patient perception of symptomatic control and adverse drug. It includes 6 scales: Symptom Interference, (4 items); Treatment Convenience, (6 items); Injection Site Interference (2 items); GI Interference (3 items); Treatment Satisfaction, (3 items); and Emotional Reaction (3 items). Each scale score can range from 0 to 100, with 0 representing the lowest (highest burden/lower satisfaction) and 100 representing the best possible score (lowest burden/highest satisfaction) for each of the 6 scales. Positive Acro-TSQ change scores indicate improvement while negative change scores indicate worsening.
Time Frame: 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 16
Participants | 0 | 13
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; This endpoint is descriptive with no formal statistical hypothesis testing; Test type: Other; The week 26 value is used as the baseline value for the RCT phase. The denominator for the percentage was the number of subjects at each visit

10. Other Pre Specified Outcome: Proportion of Patients on Octreotide Capsules Who Are Biochemically Controlled at the End of the RCT Phase- Landmark Analysis
Description: Proportion of patients on octreotide capsules who are biochemically controlled at the end of the RCT phase defined as IGF-1< 1.3 x ULN based on average of weeks 58 and 62
Time Frame: Average of weeks 58 and 62
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
Participants | 49 | 35
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; This endpoints is descriptive with no formal statistical hypothesis testing; Test type: Other; This sensitivity analysis was using the Full analysis set (FAS), where any patient who discontinued treatment early was imputed as non-responder

11. Other Pre Specified Outcome: Proportion of Week 26 Responders on Octreotide Capsules Who Are Biochemically Controlled at the End of the RCT Phase- Landmark Sensitivity Analysis
Description: Proportion of patients on Octreotide Capsules Who Are Biochemically Controlled at the End of the RCT Phase- Landmark sensitivity analysis- Week 26 responders
Time Frame: 62 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 48 | 36
Participants | 45 | 34
Statistical Analysis 1: Comparison: RCT Phase - Oral vs RCT Phase - Injectables; This endpoints is descriptive with no formal statistical hypothesis testing; Test type: Other; This sensitivity analysis was using the Full analysis set (FAS), where patient who were biochemically controlled at the RCT Baseline (week 26), and who discontinued treatment early was imputed as non-responder

12. Other Pre Specified Outcome: Proportion of Patients Biochemically Controlled at the End of Run-in
Description: Proportion of patients biochemically controlled at the end of the Run-in phase, defined as average IGF-1 levels during weeks 24 and 26 < 1.3xULN
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase
Number analyzed (Participants) | 146
Participants | 94
Statistical Analysis 1: Comparison: Run-in Phase; Test type: Other; Proportion of patients = 64.4, 95% CI 2-sided [56 to 72.1] — Confidence Interval estimated using the Clopper-Pearson (Exact) method; The proportion of patients biochemically controlled at the end of the Run-in phase was defined as IGF-1 < 1.3 times ULN [based on the average of week 24 and week 26])

13. Other Pre Specified Outcome: Proportion of Patients With a Reduction in the Overall Number of Active Acromegaly Symptoms at the End of the Run-in Phase
Description: Proportion of patients with a reduction in the overall number of active acromegaly symptoms at the end of the Run-in phase compared to Baseline
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase
Number analyzed (Participants) | 146
Participants | 97
Statistical Analysis 1: Comparison: Run-in Phase; Test type: Other; Proportion of patients = 66.4, 95% CI 2-sided [58.5 to 74.1]

14. Other Pre Specified Outcome: Proportion of Patients With Improved Acromegaly Index of Severity (AIS) Score at the End of the Run-in Phase
Description: Proportion of patients with improved AIS score at the end of the Run-in phase compared to Baseline Acromegaly index of severity (AIS) at the end of Run-in phase compared to Baseline.
  The Acromegaly Index of Severity (AIS) symptom score is calculated based on the presence and severity of 5 acromegaly signs/symptoms: headache, swelling of extremities, joint pain, sweating, and fatigue. Each symptom was graded from no symptoms (score 0), to mild symptoms (1), moderate (2), or severe symptoms (3).
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase
Number analyzed (Participants) | 92
Participants | 45
Statistical Analysis 1: Comparison: Run-in Phase; Test type: Other; Proportion of patients = 48.9, 95% CI 2-sided [38.7 to 59.1]

15. Other Pre Specified Outcome: EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) Index Scores During the Run-in Phase
Description: Change from baselines in EQ-5D-5L Index scores in randomized participants during the Run-in phase.
  EQ-5D-5L (five severity levels EQ-5D) is a standardized instrument completed by the patient for use as a measure of health outcome applicable to a wide range of health conditions. It comprises 5 dimensions of health: mobility, ability to self care, ability to undertake usual activities, pain and discomfort, and anxiety and depression. Based on qualitative and quantitative studies conducted by the EuroQol Group, there are 5 levels under each domain: 'no problems' (assigned a value of 1), 'slight problems' (assigned a value of 2), 'moderate problems' (assigned a value of 3), 'severe problems' (assigned a value of 4), and 'unable to/extreme problems' (assigned a value of 5). An EQ-5D Index score is calculated based on the responses to these 5 dimensions of health. Weights for use in the index calculation are not universally available. Higher values represent better health states.
Time Frame: 26 weeks
Population: All patients who were randomized to the RCT phase
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Run-in Phase
Number analyzed (Participants) | 92
units on a scale | 0.0433 [0.011 to 0.0755]

16. Other Pre Specified Outcome: Change From Baseline to End of RCT Phase in WPAI
Description: Work Productivity and Activity Impairment Questionnaire- RCT phase. WPAI:SHP is a standardized and validated PRO questionnaire to measure health outcomes in clinical trial settings. It measures time missed from work, impairment of work and regular activities due to overall health and symptoms, relative to measures of general health perceptions, role (physical), role (emotional), pain, symptom severity, and global measures of work and interference with regular activity.
  The WPAI yields 4 types of scores: (1) absenteeism (work time missed); (2) presenteeism (impairment at work/reduced on-the-job effectiveness); (3) work productivity loss (overall work impairment/absenteeism plus presenteeism); and (4) activity impairment. Each of the 4 WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity (i.e., worse outcomes).
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from Baseline RCT
Arm/Group | RCT Phase - Oral | RCT Phase - Injectables
Number analyzed (Participants) | 55 | 37
Percentage change from Baseline RCT
  Absenteeism (%) | -0.34 [-2.11 to 1.43] | 0.79 [-1.53 to 3.12]
  Presenteeism (%) | 1.85 [-4.48 to 8.17] | 5.98 [-2.02 to 13.98]
  Work productivity loss (%) | 1.49 [-5.09 to 8.08] | 6.93 [-1.74 to 15.59]
  Activity impairment (%) | 0.84 [-4.34 to 6.02] | 4.34 [-2.1 to 10.77]

17. Other Pre Specified Outcome: Change From Baseline to End of Run-in Phase in WPAI
Description: Work Productivity and Activity Impairment Questionnaire- Run-in phase. WPAI:SHP is a standardized and validated PRO questionnaire to measure health outcomes in clinical trial settings. It measures time missed from work, impairment of work and regular activities due to overall health and symptoms, relative to measures of general health perceptions, role (physical), role (emotional), pain, symptom severity, and global measures of work and interference with regular activity.
  The WPAI yields 4 types of scores: (1) absenteeism (work time missed); (2) presenteeism (impairment at work/reduced on-the-job effectiveness); (3) work productivity loss (overall work impairment/absenteeism plus presenteeism); and (4) activity impairment. Each of the 4 WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity (i.e., worse outcomes).
Time Frame: 62 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change from Run-in baseline
Arm/Group | Run-in Phase
Number analyzed (Participants) | 146
Percentage change from Run-in baseline
  Absenteeism (%) | -0.81 [-3.84 to 2.21]
  Presenteeism (%) | -6.65 [-12.39 to -0.9]
  Work Productivity Loss (%) | -6.92 [-12.83 to -1.02]
  Activity Impairment (%) | -4.94 [-9.17 to -0.71]

18. Other Pre Specified Outcome: Change in Acromegaly Treatment Satisfaction Questionnaire (ACRO-TSQ) Scores From Baseline to End of Run-in in Randomized Patients.
Description: Change in Acromegaly treatment satisfaction questionnaire (ACRO-TSQ) PRO questionnaire from baseline to end of Run-in phase in randomized patients.
  Acro-TSQ is a validated PRO tool assessing overall convenience and satisfaction with treatment and patient perception of symptomatic control and adverse drug. It includes 6 scales: Symptom Interference, (4 items); Treatment Convenience, (6 items); Injection Site Interference (2 items); GI Interference (3 items); Treatment Satisfaction, (3 items); and Emotional Reaction (3 items). Each scale score can range from 0 to 100, with 0 representing the lowest (highest burden/lower satisfaction) and 100 representing the best possible score (lowest burden/highest satisfaction) for each of the 6 scales. Positive Acro-TSQ change scores indicate improvement while negative change scores indicate worsening.
Time Frame: 26 weeks
Population: Change in Acro-TSQ domains in randomized patients
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Run-in Phase
Number analyzed (Participants) | 57
score on a scale
  Emotional reaction - Change from baseline | 9.65 [3.31 to 15.98]
  GI interference - Change from baseline | 4.24 [-1.32 to 9.8]
  Symptom interference- Change from baseline | 2.45 [-2.1 to 7]
  Treatment convenience - Change from baseline | 6.37 [0.25 to 12.5]
  Treatment satisfaction - Change from baseline | 6.73 [0.9 to 12.55]
Statistical Analysis 1: Comparison: Run-in Phase; Test type: Other; The LSM change from baseline estimates are from a mixed model for repeated measures

ADVERSE EVENTS:
Time Frame: 1 year, 3 months for both the Run-in and RCT phases.
Description: Safety population: All participants enrolled in the study who received any amount of the study drug.
Groups:
- Run-in Phase; RCT Phase - Oral: Oral octreotide capsules
  Octreotide capsules
- RCT Phase - Injectables: Injectable somatostatin analogs (octreotide or lanreotide)
  Octreotide capsules
- Combination Phase (Sub-study): Octreotide capsules plus cabergoline
  Octreotide capsules
Arm/Group | Run-in Phase | RCT Phase - Oral | RCT Phase - Injectables | Combination Phase (Sub-study)
All-Cause Mortality (participants affected / at risk) | 0/146 | 1/55 | 0/37 | 0/14
Serious Adverse Events (participants affected / at risk) | 6/146 | 3/55 | 3/37 | 0/14
Other Adverse Events (participants affected / at risk) | 106/146 | 39/55 | 26/37 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Phase (N=146) | RCT Phase - Oral (N=55) | RCT Phase - Injectables (N=37) | Combination Phase (Sub-study) (N=14)
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Phase (N=146) | RCT Phase - Oral (N=55) | RCT Phase - Injectables (N=37) | Combination Phase (Sub-study) (N=14)
Nausea (Gastrointestinal disorders) | 32 | 11 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 22 | 6 | 5 | 1
Flatulence (Gastrointestinal disorders) | 14 | 14 | 8 | 1
Abdominal pain (Gastrointestinal disorders) | 13 | 5 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 8 | 0 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 3 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 9 | 5 | 0 | 1
Urinary tract infection (Infections and infestations) | 8 | 2 | 0 | 0
Headache (Nervous system disorders) | 18 | 5 | 1 | 0
Dizziness (Nervous system disorders) | 9 | 0 | 3 | 0
Injection site nodule (General disorders) | 0 | 0 | 5 | 0
Injection site pain (General disorders) | 0 | 0 | 3 | 0
Peripheral swelling (General disorders) | 7 | 3 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 0
Fatigue (General disorders) | 9 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Influnza (Infections and infestations) | 0 | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT02685709/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02685709/SAP_001.pdf